CLINICAL TRIAL: NCT04339985
Title: A Randomized, Double-Blind, Parallel Group, Vehicle-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of Topical ATx201 OINTMENT in Adolescents and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: Study to Evaluate Safety & Efficacy of Topical ATx201 OINTMENT in Adolescents and Adults With Mild to Moderate AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATx201-207
Record Dates: First submitted 2020-03-23; First posted 2020-04-09 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned by using Interactive Web Response System (IWRS) to one of three treatment groups
Who Masked: Participant, Investigator
Masking Description: Approx. 210 subjects randomized and 16 subjects will be in an open-label sub-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ATx201 OINTMENT 4% (Experimental): ATx201 OINTMENT 4%
  Interventions: Drug: ATx201
- ATx201 OINTMENT 7% (Experimental): ATx201 OINTMENT 7%
  Interventions: Drug: ATx201
- ATx201 OINTMENT vehicle (Experimental): ATx201 OINTMENT vehicle
  Interventions: Drug: ATx201 OINTMENT vehicle

INTERVENTIONS:
Drug: ATx201 — Topical
  Other Names: ATx201 OINTMENT
  Arms: ATx201 OINTMENT 4%; ATx201 OINTMENT 7%
Drug: ATx201 OINTMENT vehicle — ATx201 OINTMENT vehicle
  Arms: ATx201 OINTMENT vehicle

SUMMARY:
This is a Phase 2 randomized, double-blind, parallel group, vehicle-controlled study to evaluate the safety and efficacy of topical ATx201 OINTMENT in adolescents and adults with mild to moderate Atopic Dermatitis

DETAILED DESCRIPTION:
This is a Phase 2 randomized, double-blind, parallel group, vehicle-controlled study to evaluate the safety and efficacy of topical ATx201 OINTMENT in adolescents and adults with mild to moderate Atopic Dermatitis.

Approximately 210 subjects will be randomly assigned to receive ATx201 OINTMENT 4%, ATx201 OINTMENT 7%, or OINTMENT vehicle for 6 weeks. Treatments will be balanced into consecutive blocks in 1:1:1 ratio for the active groups and vehicle.

Sixteen additional subjects (adults and adolescents) will be enrolled in a 2-week open label substudy of twice-daily ATx201 OINTMENT 7% to evaluate the PK profile of ATx201.

ELIGIBILITY:
Inclusion Criteria (main ones):

1. Diagnosis of AD using the Hanifin and Rajka criteria and minimum 1-year history with a current IGA score of 2 or 3 and treatable BSA ≥5% but ≤36% (treatable BSA includes all lesions present at screening except scalp)
2. Age ≥12 and <60 years
3. Male or nonpregnant and nonlactating female who is abstinent or agrees to use effective contraceptive methods throughout the course of the study. Females must have a negative urine beta-human chorionic gonadotropin hormone (hCG) pregnancy test at Day 1.
4. Subject or LAR able to understand and provide signed informed consent. Assent is also required of adolescents.
5. Normally active and otherwise in good health by medical history and physical examination

Exclusion Criteria (main ones):

1. Actively infected AD (ie, requiring antimicrobial therapy as determined by the investigator)
2. Acute exacerbation or flare in the 4 weeks prior to the Day 1 visit that necessitates treatment with a high potency corticosteroid (such as clobetasol propionate or betamethasone dipropionate), or antibiotics, or prednisolone
3. Enrollment in an ATx201 study in the previous 6 months
4. Allergy or history of significant adverse reaction to ATx201 or related compounds, or to any of the excipients used
5. Underlying skin condition that may interfere with the placement of study treatment or impede clinical evaluations (including active Herpes simplex)
6. Current acute or chronic condition unless considered clinically irrelevant and stable by the investigator
7. The presence of a condition the investigator believes would interfere with the ability to provide informed consent or assent, or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk
8. Unable or unwilling to comply with study procedures
9. Exposure to any IP within 30 days prior to randomization

There are also some specific criteria related to prior or concomitant therapy

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline at Week 6 in Eczema Area Severity Index (EASI) | Baseline to Week 6
  EASI mean change from baseline at Week 6

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) success | Baseline to Week 6
  IGA success with defined improvement from baseline; success defined as clear (0) or almost clear (1) with ≥2 grade improvement from baseline
change from baseline in Investigator Global Assessment (IGA) scoring | Baseline to Week 6
  Distribution of IGA scores and change from baseline
Mean change from baseline in Target lesion Total Sign Score (TSS) | Baseline to Week 6
  Target lesion TSS mean change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Andres, Dr., Study Chair — UNION therapeutics
Locations (10):
- Bulgaria (4):
  - UNION therapeutics Investigational Site 5, Pleven
  - UNION therapeutics Investigational Site 2, Sofia
  - UNION therapeutics Investigational Site 3, Sofia
  - UNION therapeutics Investigational Site 4, Sofia
- UNION therapeutics Investigational Site 1, Herlev, Denmark
- Poland (5):
  - UNION therapeutics Investigational Site 6, Bydgoszcz
  - UNION therapeutics Investigational Site 10, Lodz
  - UNION therapeutics Investigational Site 7, Nowy Targ
  - UNION therapeutics Investigational Site 9, Skierniewice
  - UNION therapeutics Investigational Site 8, Wroclaw

IPD SHARING:
Plan to Share IPD: No